CLINICAL TRIAL: NCT04682366
Title: Evaluating the Effect of Tamsulosin on Postoperative Urinary Retention in Women Undergoing Same Day Hospital Discharge Following Pelvic Reconstructive Surgery: A Randomized Trial
Brief Title: The Effect of Tamsulosin on Postoperative Urinary Retention
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Challenges in enrollment led to decission for termination
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00070462
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Results first posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2022-10

CONDITIONS: Urinary Retention
Keywords: Postoperative care; Urinary tract infection; Female pelvic reconstructive surgery; Enhanced recovery after surgery; Tamsulosin; Flomax
MeSH Terms: conditions — Urinary Retention; Urinary Tract Infections | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tamsulosin (Experimental): Patients in this arm will receive 10 days of 0.4 mg of oral tamsulosin once daily starting 5 days pre-operatively and continuing until all pills are completed.
  Interventions: Drug: Tamsulosin
- Placebo (Placebo Comparator): Patients in this arm will receive 10 days of identical-appearing placebo once daily starting 5 days pre-operatively and continuing until all pills are completed.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamsulosin — Oral drug: 10 days of 0.4 mg of oral Tamsulosin
  Arms: Tamsulosin
Drug: Placebo — Oral drug: 10 days of identical-appearing placebo
  Arms: Placebo

SUMMARY:
This is a double-blinded randomized controlled trial of perioperative use of tamsulosin to prevent postoperative urinary retention in female pelvic reconstructive surgery undergoing same-day discharge with an enhanced recovery after surgery protocol.

DETAILED DESCRIPTION:
The primary objective is to determine the effect of Tamsulosin on same-day active voiding trial in women undergoing female pelvic reconstructive surgery with vaginal native tissue repair with same-day discharge planned.

Duration of catheterization, postoperative urinary tract infection rates, patient level of satisfaction, Emergency Department (ED) visits and adverse events postoperatively will also be compared between women receiving Tamsulosin versus placebo.

Patients will be offered participation in the study at their postoperative visit if they meet study criteria. Once consent is obtained, patients will be randomized to receive Tamsulosin 0.4 mg orally once daily or matching placebo capsules for a total of 10 days starting 5 days pre-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Stage II or greater pelvic organ prolapse in > 1 vaginal compartment
* Plan for multicompartment native tissue vaginal repair (which would include any combination of uterosacral ligament suspension, sacrospinous ligament suspension, cystocele and/or rectocele repair, with or without hysterectomy and with or without concomitant mid-urethral sling) or vaginal closure with female pelvic medicine and reconstructive surgery (FPMRS) - trained surgeons at Wake Forest Baptist Health
* Participation in Enhanced-Recovery-After-Surgery protocol with plan for same-day hospital discharge
* Willing to remain compliant with Investigation Product (IP)

Exclusion Criteria:

* Intraoperative complication necessitating prolonged bladder drainage or placement of a vaginal pack x 24 hours (patients would exit study after randomization and will be excluded from the per-protocol analysis)
* Patients whose surgical plan would necessitate a voiding trial on postop day >0
* Less than 21 years of age
* Unable to understand English
* Patients who are scheduled to undergo combined colorectal procedures such as rectopexy, sphincteroplasty
* Patient with known allergy to Tamsulosin or sulfa drugs
* Patients with upcoming cataract surgery
* Patient with orthostatic hypotension
* History of postvoid residual (PVR>150) prior to surgery with prolapse reduction
* Patients with hypertension on alpha-blockers
* Single compartment prolapse repair (anterior or posterior repair only)
* Use of mesh for prolapse repair
* High tone pelvic floor dysfunction

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 4 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Majid Mirzazadeh, MD, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Committee Opinion No 701: Choosing the Route of Hysterectomy for Benign Disease. Obstet Gynecol. 2017 Jun;129(6):e155-e159. doi: 10.1097/AOG.0000000000002112. PMID 28538495
- [Background] Akkoc A, Aydin C, Topaktas R, Kartalmis M, Altin S, Isen K, Metin A. Prophylactic effects of alpha-blockers, Tamsulosin and Alfuzosin, on postoperative urinary retention in male patients undergoing urologic surgery under spinal anaesthesia. Int Braz J Urol. 2016 May-Jun;42(3):578-84. doi: 10.1590/S1677-5538.IBJU.2015.0256. PMID 27286124
- [Background] Carter-Brooks CM, Du AL, Ruppert KM, Romanova AL, Zyczynski HM. Implementation of a urogynecology-specific enhanced recovery after surgery (ERAS) pathway. Am J Obstet Gynecol. 2018 Nov;219(5):495.e1-495.e10. doi: 10.1016/j.ajog.2018.06.009. Epub 2018 Jun 18. PMID 29913175
- [Background] Chapman GC, Sheyn D, Petrikovets A, Mahajan ST, El-Nashar S, Pollard R, Mangel JM. Tamsulosin to Prevent Postoperative Urinary Retention After Female Pelvic Reconstructive Surgery. Female Pelvic Med Reconstr Surg. 2020 Nov;26(11):682-687. doi: 10.1097/SPV.0000000000000650. PMID 30418263
- [Background] Chong C, Kim HS, Suh DH, Jee BC. Risk factors for urinary retention after vaginal hysterectomy for pelvic organ prolapse. Obstet Gynecol Sci. 2016 Mar;59(2):137-43. doi: 10.5468/ogs.2016.59.2.137. Epub 2016 Mar 16. PMID 27004205
- [Background] Clancy C, Coffey JC, O'Riordain MG, Burke JP. A meta-analysis of the efficacy of prophylactic alpha-blockade for the prevention of urinary retention following primary unilateral inguinal hernia repair. Am J Surg. 2018 Aug;216(2):337-341. doi: 10.1016/j.amjsurg.2017.02.017. Epub 2017 Mar 14. PMID 28341140
- [Background] Costantini E, Lazzeri M, Bini V, Zucchi A, Fioretti F, Frumenzio E, Porena M. Open-label, longitudinal study of tamsulosin for functional bladder outlet obstruction in women. Urol Int. 2009;83(3):311-5. doi: 10.1159/000241674. Epub 2009 Oct 13. PMID 19829032
- [Background] Doll KM, Dusetzina SB, Robinson W. Trends in Inpatient and Outpatient Hysterectomy and Oophorectomy Rates Among Commercially Insured Women in the United States, 2000-2014. JAMA Surg. 2016 Sep 1;151(9):876-7. doi: 10.1001/jamasurg.2016.0804. No abstract available. PMID 27168235
- [Background] FitzGerald MP, Brubaker L. The etiology of urinary retention after surgery for genuine stress incontinence. Neurourol Urodyn. 2001;20(1):13-21. doi: 10.1002/1520-6777(2001)20:13.0.co;2-r. PMID 11135378
- [Background] Geynisman-Tan J, Dave-Heliker B, Bochenska K, Collins S, Lewicky-Gaupp C, Mueller M, Kenton K. Duration of Catheterization After Retropubic Midurethral Sling. Female Pelvic Med Reconstr Surg. 2019 Sep-Oct;25(5):369-371. doi: 10.1097/SPV.0000000000000569. PMID 29509646
- [Background] Hooton TM, Bradley SF, Cardenas DD, Colgan R, Geerlings SE, Rice JC, Saint S, Schaeffer AJ, Tambayh PA, Tenke P, Nicolle LE; Infectious Diseases Society of America. Diagnosis, prevention, and treatment of catheter-associated urinary tract infection in adults: 2009 International Clinical Practice Guidelines from the Infectious Diseases Society of America. Clin Infect Dis. 2010 Mar 1;50(5):625-63. doi: 10.1086/650482. PMID 20175247
- [Background] Jackson J, Davies P, Leggett N, Nugawela MD, Scott LJ, Leach V, Richards A, Blacker A, Abrams P, Sharma J, Donovan J, Whiting P. Systematic review of interventions for the prevention and treatment of postoperative urinary retention. BJS Open. 2018 Nov 19;3(1):11-23. doi: 10.1002/bjs5.50114. eCollection 2019 Feb. PMID 30734011
- [Background] Jennings AJ, Spencer RJ, Medlin E, Rice LW, Uppal S. Predictors of 30-day readmission and impact of same-day discharge in laparoscopic hysterectomy. Am J Obstet Gynecol. 2015 Sep;213(3):344.e1-7. doi: 10.1016/j.ajog.2015.05.014. Epub 2015 May 14. PMID 25981843
- [Background] Kenton K, Pham T, Mueller E, Brubaker L. Patient preparedness: an important predictor of surgical outcome. Am J Obstet Gynecol. 2007 Dec;197(6):654.e1-6. doi: 10.1016/j.ajog.2007.08.059. PMID 18060968
- [Background] Kowalik U, Plante MK. Urinary Retention in Surgical Patients. Surg Clin North Am. 2016 Jun;96(3):453-67. doi: 10.1016/j.suc.2016.02.004. PMID 27261788
- [Background] Koyanagi T, Morita H, Taniguchi K, Kubota M, Shinno Y, Takamatsu T. Neurogenic urethra: clinical relevance of isolated neuropathic dysfunction of the urethra, and the denervation supersensitivity of the urethra revisited. Eur Urol. 1988;15(1-2):77-83. doi: 10.1159/000473401. PMID 2850917
- [Background] Livne PM, Kaplan B, Ovadia Y, Servadio C. Prevention of post-hysterectomy urinary retention by alpha-adrenergic blocker. Acta Obstet Gynecol Scand. 1983;62(4):337-40. doi: 10.3109/00016348309156234. PMID 6138916
- [Background] Lose G, Lindholm P. Prophylactic phenoxybenzamine in the prevention of postoperative retention of urine after vaginal repair: a prospective randomized double-blind trial. Int J Gynaecol Obstet. 1985 Sep;23(4):315-20. doi: 10.1016/0020-7292(85)90026-8. PMID 2866119
- [Background] Madani AH, Aval HB, Mokhtari G, Nasseh H, Esmaeili S, Shakiba M, Shakiba RS, Seyed Damavand SM. Effectiveness of tamsulosin in prevention of post-operative urinary retention: a randomized double-blind placebo-controlled study. Int Braz J Urol. 2014 Jan-Feb;40(1):30-6. doi: 10.1590/S1677-5538.IBJU.2014.01.05. PMID 24642148
- [Background] Perron-Burdick M, Yamamoto M, Zaritsky E. Same-day discharge after laparoscopic hysterectomy. Obstet Gynecol. 2011 May;117(5):1136-1141. doi: 10.1097/AOG.0b013e318215dd4e. PMID 21508753
- [Background] Poylin V, Curran T, Cataldo T, Nagle D. Perioperative use of tamsulosin significantly decreases rates of urinary retention in men undergoing pelvic surgery. Int J Colorectal Dis. 2015 Sep;30(9):1223-8. doi: 10.1007/s00384-015-2294-7. Epub 2015 Jun 23. PMID 26099320
- [Background] Propst K, Tunitsky-Bitton E, O'Sullivan DM, Steinberg AC, LaSala C. Phenazopyridine for Evaluation of Ureteral Patency: A Randomized Controlled Trial. Obstet Gynecol. 2016 Aug;128(2):348-355. doi: 10.1097/AOG.0000000000001472. PMID 27399998
- [Background] Pummangura N, Kochakarn W. Efficacy of tamsulosin in the treatment of lower urinary tract symptoms (LUTS) in women. Asian J Surg. 2007 Apr;30(2):131-7. doi: 10.1016/S1015-9584(09)60146-9. PMID 17475584
- [Background] Reitz A, Haferkamp A, Kyburz T, Knapp PA, Wefer B, Schurch B. The effect of tamsulosin on the resting tone and the contractile behaviour of the female urethra: a functional urodynamic study in healthy women. Eur Urol. 2004 Aug;46(2):235-40; discussion 240. doi: 10.1016/j.eururo.2004.04.009. PMID 15245819
- [Background] Ripperda CM, Kowalski JT, Chaudhry ZQ, Mahal AS, Lanzer J, Noor N, Good MM, Hynan LS, Jeppson PC, Rahn DD. Predictors of early postoperative voiding dysfunction and other complications following a midurethral sling. Am J Obstet Gynecol. 2016 Nov;215(5):656.e1-656.e6. doi: 10.1016/j.ajog.2016.06.010. Epub 2016 Jun 16. PMID 27319367
- [Background] Schiavone MB, Herzog TJ, Ananth CV, Wilde ET, Lewin SN, Burke WM, Lu YS, Neugut AI, Hershman DL, Wright JD. Feasibility and economic impact of same-day discharge for women who undergo laparoscopic hysterectomy. Am J Obstet Gynecol. 2012 Nov;207(5):382.e1-9. doi: 10.1016/j.ajog.2012.09.014. Epub 2012 Sep 17. PMID 23107080
- [Background] Tunitsky-Bitton E, Murphy A, Barber MD, Goldman HB, Vasavada S, Jelovsek JE. Assessment of voiding after sling: a randomized trial of 2 methods of postoperative catheter management after midurethral sling surgery for stress urinary incontinence in women. Am J Obstet Gynecol. 2015 May;212(5):597.e1-9. doi: 10.1016/j.ajog.2014.11.033. Epub 2014 Nov 27. PMID 25434837
- [Background] Turner LC, Kantartzis K, Shepherd JP. Predictors of postoperative acute urinary retention in women undergoing minimally invasive sacral colpopexy. Female Pelvic Med Reconstr Surg. 2015 Jan-Feb;21(1):39-42. doi: 10.1097/SPV.0000000000000110. PMID 25185611

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tamsulosin | Placebo
Started | 2 | 2
Completed | 1 | 1
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: 2 Subjects were Lost To Follow - 1 in each Group
Groups:
- Total: Total of all reporting groups
Arm/Group | Tamsulosin | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants] — Population: 1 Subject was Lost-to-Follow
  Participants
    number analyzed (Participants) | 1 | 1 | 2
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 Subject in each group was LTF
  Participants
    number analyzed (Participants) | 1 | 1 | 2
    Female | 1 | 1 | 2
    Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 1 Subject in each group was LTF
  Participants
    number analyzed (Participants) | 1 | 1 | 2
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 1 | 1 | 2
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2
Lost to follow-up [Count of Participants; unit: Participants] | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative (Day 0) Urinary Retention
Description: Urinary retention can be defined as >150cc residual volume during an active voiding trial
Time Frame: Up to 6 weeks postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

2. Secondary Outcome: Urinary Tract Infection Rate
Description: Urinary tract infection rate
Time Frame: Week 6
Population: No Data was collected
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Incidence of Delayed Urinary Retention
Description: Delayed urinary retention will be defined as post-void residual > 150 cc
Time Frame: Week 6
Population: No Data was collected
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number Emergency Department (ED) Visits
Time Frame: Up to 30 days postoperatively
Population: No Data was collected
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Total Number of Days of Bladder Catheterization
Time Frame: Week 6
Population: No Data was collected
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Patient Level of Satisfaction With Voiding Function
Description: Patient satisfaction questionnaire: Patient Global Impression of Improvement (PGI-I) - Patient level of satisfaction (scale of 1 -7) - very dissatisfied, moderately dissatisfied, slightly dissatisfied, neutral, slightly satisfied, moderately satisfied, very satisfied - the lower the score denotes the more satisfaction)
Time Frame: Day 0 and 1 week postoperatively
Population: No Data was collected
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Tamsulosin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 0/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tamsulosin (N=1) | Placebo (N=1)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT04682366/Prot_SAP_003.pdf
  • Informed Consent Form (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT04682366/ICF_000.pdf